CLINICAL TRIAL: NCT06749873
Title: Assessing Helicobacter Pylori Diagnosis and Treatment Quality of direct-to Consumer Telemedicine in Mainland China: a Cross-sectional Study Using Unannounced Standardised Patients
Brief Title: Assessing Hp Diagnosis and Treatment Quality of direct-to Consumer Telemedicine in Mainland China
Acronym: Hp
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Professor, Shandong University
Other Study IDs: QLYY-2024-001; 82270570 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2024-11-30; First posted 2024-12-27 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Sp was asked with the following baseline information: 1. 20 years of age and gender; 2. positive urea breath test; 3. no symptoms; 4. no family history of gastric cancer; 5. gastroscopy: non-atrophic gastritis; 6. no treatments; and 7. no history of drug allergies.
  Interventions: Other: Background of different SP information

INTERVENTIONS:
Other: Background of different SP information — Sp was asked with the following baseline information: 1. 50 years of age and gender; 2. positive urea breath test; 3. asymptomatic; 4. family history of gastric cancer; 5. gastroscopy: atrophic gastritis; 6. untreated; and 7. no history of drug allergies.

SUMMARY:
A quality assessment of the level of H. pylori diagnosis and treatment in mainland China's Direct-to-consumer telemedicine (DTCT) was conducted by means of Unannounced standardized patients (USPs).

DETAILED DESCRIPTION:
Direct-to-consumer telemedicine (DTCT) refers to a model in which doctors provide medical advice and services directly to patients through the Internet and communication technologies. Under the background of globalization and information age, DTCT, as an innovative medical service model, is gradually changing the traditional face of the medical industry. Especially in today's highly developed information and network, telemedicine service has become an important way to improve the accessibility of medical services, reduce medical costs, and optimize the allocation of medical resources. In China, with the in-depth implementation of the Healthy China strategy, DTCT is regarded as a key link to deepen medical reform and build a new medical service system. In 2018, the Chinese government began to introduce a series of DTCT policy measures to promote the development of telemedicine. By June 2022, China has approved and set up more than 1,700 Internet hospitals, initially forming an integrated online and offline medical services2. As of February 2024, China's National Health Commission has approved the establishment of more than 2,700 Internet hospitals across the country. In addition to the Internet hospitals dominated by physical hospitals, the enterprise-led Internet medical consulting platform has also gradually flourished and gradually occupied a large market share.

The speed of development of DTCT is encouraging, but the quality of care in DTCT is more uncertain. In 2024, a Chinese study published was the first to evaluate multi-disease online diagnosis and treatment services offered on Chinese Internet diagnosis and treatment platforms, using anonymous standardized patients. The study found that the current quality of Internet diagnosis and treatment services is not ideal: out of 170 anonymous consultations, the access success rate is only 63.5% (108/170); Of the visits successfully completed, only 49 consultations (45%) resulted in a correct diagnosis. In terms of physician adherence to the guidelines, the rate of completion of consultation and disposal was 15% and 31%, respectively.

Helicobacter pylori (Hp) infection is a common gastrointestinal disease, which is closely related to the occurrence of gastritis, peptic ulcer, gastric cancer and other diseases. Globally, 43.1% of the population is infected with Helicobacter pylori. In China, the infection rate is also close to 50%. Hp infection has a huge demand for treatment, and it also faces many problems such as complicated treatment plan. Direct-to-consumer telemedicine services offer new possibilities for the treatment of Hp infection, greatly facilitating patients, especially those in remote areas and primary care facilities. However, there is uncertainty in the quality of H. pylori treatment in telemedicine services.

ELIGIBILITY:
Inclusion Criteria:

* An Internet hospital dominated by physical hospitals in the seven geographical regions of gastroenterology specialty reputation shortlisted by the Hospital Research Institute of Fudan University in China
* Be included in the top 20 enterprise-led Internet medical consulting platforms based on popularity and user recognition

Exclusion Criteria:

* Physical hospitals without Internet hospitals
* The entity hospital of the Internet hospital can only be revisited

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Undeclared Standardized patient (USP) usually refers to a teaching tool used in medical education and training. These standardized patients are trained actors who simulate the conditions, symptoms, and emotional responses of real patients to help physicians improve their clinical skills. In the "undeclared" scenario, these standardized patients may not reveal their identity at the outset, but participate in training or evaluation as real patients, allowing medicine to diagnose and treat without prior preparation. This approach can more realistically simulate the clinical environment and help improve clinical thinking skills, communication skills and understanding of patients.
  It is expected that 10 research assistants will be included for USP training.
Sampling Method: Non-Probability Sample
Enrollment: 552 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Guidelines compliance | 3 months
  For the doctor's inquiry through SP, the doctor's answer will be scored against the current guidelines, and the correct answer according to the guidelines will get the corresponding score, out of 10 points. Adherence to the physician's guidelines will be judged by the high or low scores assessed.
Patient satisfaction | 3 months
  Through the SP for the doctor's inquiry, the doctor's attitude will be scored, and the corresponding score will be obtained. The patient's satisfaction with the physician will be judged by the high or low score of the assessment

SECONDARY OUTCOMES:
Response rate | 3 months
  Ratio of physician responses to consultations in Internet hospitals

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandoang, China